CLINICAL TRIAL: NCT06005363
Title: The Application of Anesthesia Depth Monitoring on Post-operative Cognitive Dysfunction for Patients With Hydrocephalus Receiving Ventricular-peritoneal Shunt Surgery and Associated Change in CSF Metabolomics and Glymphatic Function.
Brief Title: CSF Metabolomics and Glymphatic Function in Patients Receiving VP- Shunt Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CMRPG3N0591
Record Dates: First submitted 2023-08-07; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: The Association of Postoperative Cognitive Dysfunction With Glymphatic Function and Neuroinflammation; The Association of Postoperative Cognitive Dysfunction With CSF Metabolomic Change
Keywords: anesthesia depth monitoring; postoperative cognitive dysfunction; metabolomics; cerebrospinal fluid; glymphatic function
MeSH Terms: conditions — Neuroinflammatory Diseases; Postoperative Cognitive Complications | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Two interventional group with BIS group and DEX group all receive BIS monitoring, and DEX group receive dexmedetomidine infusion.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants receive randomized allocation to BIS, DEX, or usual care group before VP shunt surgery. Outcome assessor evaluate the preoperative and postoperative cognitive function, delirium status, and evaluate glymphatic function with functional MRI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIS group (Experimental): Use BIS monitoring to adjust intraoperative anesthetics.
  Interventions: Device: anesthesia depth monitoring
- DEX group (Experimental): use BIS monitoring to adjust anesthetics and give dexmedetomidine infusion.
  Interventions: Drug: Dexmedetomidine; Device: anesthesia depth monitoring
- Usual group (No Intervention): usual care with 1 MAC sevoflurane maintainance.

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine infusion
  Other Names: DEX
  Arms: DEX group
Device: anesthesia depth monitoring — intraoperative anesthesia depth monitoring to keep BIS 40-60
  Other Names: BIS
  Arms: BIS group; DEX group

SUMMARY:
In this randomized control study, the investigators intended to evaluate the influence of different anesthetics on postoperative cognitive dysfunction, neuroinflammation, CSF metabolomics, and glymphatic function in patients with normal pressure hydrocephalus for VP shunt surgery. The investigators assume that the use of dexmedetomidine infusion and proper anesthsia depth during general anesthesia, in addition to multi-model analgesia, might be helpful to enhance glymphatic function, reduce neuroinflammation, and decrease postoperative cognitive dysfunction.

DETAILED DESCRIPTION:
In this prospective randomized controlled study, 48 patients with communicating hydrocephalus will be enrolled in the study and these patients will be divided into 3 groups in which intervention group received anesthesia depth monitoring (BIS group and DEX group) and dexmedetomidine infusion (DEX group), while the controlled group received usual anesthesia care without dexmedetomidine during VP shunt surgery. The participant's intraoperative CSF and plasma samples will be collected for biochemical analysis and metabolomic analysis. The investigators will use two analytical metabolomic platforms, including nuclear magnetic resonance (NMR) and liquid chromatography-mass spectrometry (LC-MS), to execute quantitative metabolomics on human CSF and plasma samples. These metabolomic data will be compared with previous established human aging CSF Metabolome Database. After VP shunt surgery, these patient's glymphatic function will be evaluated with 3T functional MRI. The postoperative cognitive function and delirium status of these patients will be evaluated for the following 3 days using MMSE score, Montreal Cognitive Assessment, and CAM-ICU score. During analysis, the pre-operative metabolomic signature of patients with postoperative cognitive dysfunction(POCD) will be compared with patients without POCD to profile the metabolomics of POCD. Besides, the investigators could examine the correlation of glymphatic function and POCD. By comparing the CSF metabolomic change in these three groups, the investigators could evaluate the the efficacy of anesthesia depth monitoring and dexmedetomidine to reduce POCD development during VP shunt surgery. The result of this study might be able to explain the brain pathophysiology of POCD, the role of glymphatic function in POCD, metabolomic signature of POCD, and establish a better anesthesia regimen to reduce the development of POCD.

ELIGIBILITY:
Inclusion Criteria:

* patients with communicating hydrocephalus for elective VP shunt surgery under general anesthesia
* age> 60 y/o
* conscious clear
* fluency in Chinese
* anticipated hospital stay ≥ 3 days after surgery

Exclusion Criteria:

* unstable preoperative condition (unstable angina, CHF, asthma attack) within 4 weeks before surgery,
* severe hepatic dysfunction or renal failure
* history of neuropsychological diseases such as schizophrenia, Parkinson's disease, dementia, stroke,
* pre-op cognitive impairment,
* preoperative delirium,
* preoperative depression,
* allergy to contrast medium of MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative cognitive function | postoperative 2 hours, postoperative day 1, postoperative day 2, postoperative day 3
  MMSE, MoCA, CAM-ICU score
NMR amd LC-MS CSF and plasma metabolomics | preoperative, postoperative 2 hours, postoperative day 1
  NMR and LC-MS metabolomics of CSF and plasma samples

SECONDARY OUTCOMES:
Neuroinflammation parameters | preoperative, postoperative 2 hours, postoperative day 1
  lactate, tau protein, amyloid beta, orexin, IL-6, IL-10, TNF-alpha, s100b
Glymphatic function | preoperative, postoperative day 1
  evaluate DTI-ALPS index in 3T functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Huan-tang Lin, Principal Investigator — Department of anesthesiology, Linkou Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
personal data is encrypted